CLINICAL TRIAL: NCT06285058
Title: A Artificial Intelligence Model Predicts Pathological Complete Response of Lung Cancer Following Neoadjuvant Immunochemotherapy
Brief Title: Deep Learning Model Predicts Pathological Complete Response of Lung Cancer Following Neoadjuvant Immunochemotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: LUNAI
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Deep Learning Model; Pathological Complete Response; Non-small Cell Lung Cancer; Neoadjuvant Chemoimmunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training dataset: patients who were diagnosed with non-small cell carcinoma and undergo surgery after neoadjuvant chemoimmunotherapy treatment at hospital 1 (Tongji Medical College Affiliated Union Hospital)
  Interventions: Diagnostic Test: No interventions
- test dataset: patients who were diagnosed with non-small cell carcinoma and undergo surgery after neoadjuvant chemoimmunotherapy treatment at hospital (Zhengzhou University First Affiliated Hospital, Yichang Central Hospital, Anyang Cancer Hospital)

INTERVENTIONS:
Diagnostic Test: No interventions — The high-throughput extraction of large amounts of quantitative image features from medical images
  Groups: Training dataset

SUMMARY:
This study presents the development and validation of an artificial intelligence (AI) prediction system that utilizes pre-neoadjuvant immunotherapy plain scans and enhanced multimodal CT scans to extract deep learning features. The aim is to predict the occurrence of pathological complete response in non-small cell lung cancer patients undergoing neoadjuvant immunochemotherapyy.

DETAILED DESCRIPTION:
This study retrospectively obtained non-contrast enhanced and contrast enhanced CT scans of patients with NSCLC who underwent surgery after receiving neoadjuvant immunochemotherapy. at multiple centers between August 2019 and February 2023. Deep learning features were extracted from both non-contract enhanced and contract enhanced CT scans to construct the predictive models (LUNAI-nCT model and LUNAI-eCT model), respectively. After feature fusion of these two types of features, a fused model (LUNAI-fCT model) was constructed. The performance of the model was evaluated using the area under the receiver operating characteristic curve (AUC), accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV). SHapley Additive exPlanations (SHAP) analysis was used to quantify the impact of CT imaging features on model prediction. To gain insights into how our model makes predictions, we employed Gradient-weighted Class Activation Mapping (Grad-CAM) to generate saliency heatmaps.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' with non-small cell lung cancer, diagnosed through biopsy pathology and clinically classified as stage IB to III;
2. Patients who receive at least two cycles of neoadjuvant immunotherapy combined with chemotherapy induction therapy;
3. According to the IASLC guidelines, postoperative pathological evaluation was performed on the treatment response of the tumor primary lesion and lymph nodes.

Exclusion Criteria:

1. Missing or inadequate quality of CT;
2. Time interval between CT and start of treatment is greater than 1 month;
3. Incomplete clinicopathologic data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were diagnosed with non-small cell carcinoma and undergo surgery after neoadjuvant chemoimmunotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
the accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of predicting model | Baseline treatment
  several metrics were calculated, including accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ye G, Wei Z, Han C, Wu G, Wong C, Liang Y, Chen X, Zhou W, Gao J, Liang C, Liao Y, Hendriks LEL, Wee L, De Ruysscher D, Dekker A, Zhou H, Qi Y, Liu Z, Shi Z. AI-derived longitudinal and multi-dimensional CT classifier for non-small cell lung cancer to optimize neoadjuvant chemoimmunotherapy decision: a multicentre retrospective study. EClinicalMedicine. 2025 Oct 7;89:103551. doi: 10.1016/j.eclinm.2025.103551. eCollection 2025 Nov. PMID 41127561